CLINICAL TRIAL: NCT06908434
Title: A Phase I, Multicenter, Multinational, Open-label, First-in-Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of GenSci128 Tablet in Patients With Locally Advanced or Metastatic Solid Tumors Harboring a TP53 Y220C Mutation
Brief Title: A Phase I First-in-Human Study of GenSci128 in Patients With Solid Tumors Harboring a TP53 Y220C Mutation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GenSci128-101
Record Dates: First submitted 2025-03-19; First posted 2025-04-03 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumors Harboring a TP53 Y220C Mutation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 150mg dose level (Experimental)
  Interventions: Drug: GenSci128 tablets
- 300mg dose level (Experimental)
  Interventions: Drug: GenSci128 tablets
- 600mg dose level (Experimental)
  Interventions: Drug: GenSci128 tablets
- 1200mg dose level (Experimental)
  Interventions: Drug: GenSci128 tablets
- 1800mg dose level (Experimental)
  Interventions: Drug: GenSci128 tablets
- 2500mg dose level (Experimental)
  Interventions: Drug: GenSci128 tablets

INTERVENTIONS:
Drug: GenSci128 tablets — GenSci128 tablets have three specifications, including 50mg, 200mg, 500mg, and are taken in combination with the doctor's advice in different dose levels. GenSci128 will be orally administrated daily (except single dose in Cycle 0) with no interruptions until occurrence of unacceptable toxicity, or progressive disease, or withdrawal of consent, or death, or contact lost, or starting a new anticancer therapy, etc. (whichever occurs first).

SUMMARY:
The purpose of this study is to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of GenSci128 Tablet in Patients with Locally Advanced or Metastatic Solid Tumors Harboring a TP53 Y220C Mutation

ELIGIBILITY:
Inclusion Criteria:

1. Has the ability to understand and the willingness to sign a written informed consent document (prior to the initiation dose of GenSci128 and any study procedures)
2. Is willing and able to comply with the scheduled visits, treatment plan, laboratory tests and other specified study procedures
3. Has confirmed TP53 Y220C mutation in tumor tissue
4. Has histologically or cytologically confirmed locally advanced or metastatic solid tumors and have progressed following standard therapy, or for whom, in the opinion of the investigator, no available and effective standard therapy exists.
5. Has at least one measurable lesion by RECIST v1.1
6. Has an ECOG status of 0 or 1
7. Has a life expectancy of ≥ 3 months.

Exclusion Criteria:

1. Has diagnosed as primary central nervous system (CNS) tumor.
2. Has CNS metastases, unless asymptomatic, neurologically stable and not requiring steroids treatment for at least 2 weeks prior to initiation dose of GenSci128.
3. Has a history of leptomeningeal disease or spinal cord compression.
4. Has stroke or transient ischemic attack within 6 months prior to initiation dose of GenSci128.
5. Has active infection requiring intravenous (IV) antibiotics or other uncontrolled inter-current illness requiring hospitalization. Minor infections, e.g., periodontal infection or urinary tract infection (UTI), which may be treated with short term oral antibiotics are allowed.
6. Uncontrolled hypertension (Blood pressure ≥ 150/90 mmHg despite optimal medical management)
7. Has a history of prior organ transplant or allogeneic stem cell transplant.
8. Has received a selective reactivator of p53 Y220C mutation.
9. Has uncontrollable pleural effusion, pericardial effusion, or ascites requiring frequent drainage (recurrence ≤ 14 days after intervention).
10. Has known human immunodeficiency virus (HIV) infection (positive HIV 1/2 antibodies) or known chronic hepatitis B or C [participants positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) will be eligible if they are negative for HBV-DNA; participants positive for hepatitis C virus (HCV) IgG will be eligible if they are negative for HCV-RNA].
11. Is persisting toxicity related to prior anticancer therapy (NCI CTCAE V5.0 Grade>1). However, alopecia and sensory neuropathy Grade ≤2, or other Grade ≤2 adverse events not constituting a safety risk, based on the investigator's judgment are acceptable.
12. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or GenSci128 administration or may interfere with the interpretation of study results, in the judgment of the investigator, would make the participant inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) and dose limiting toxicities (DLTs) | 3 weeks
  Part 1 is a dose escalation study ，to assess the safety and tolerability of GenSci128 in participants with locally advanced or metastatic solid tumors harboring a TP53 Y220C mutation
maximal tolerance dose （MTD）、recommended dose of expansion （RDE） | up to 3 months
  Part 1 is a dose escalation study ，to determine the maximum tolerated dose (MTD), if any, and recommend dose of expansion (RDE) for GenSci128 in participants with locally advanced or metastatic solid tumors harboring a TP53 Y220C mutation
recommended phase 2 dose （RP2D） | up to 3 months
  Part 2 is a dose expansion study，Determining Recommended Phase II Dose

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital ,Fudan University, Shanghai, Shanghai Municipality, China